CLINICAL TRIAL: NCT07389252
Title: Effectiveness of Fascial Manipulation on Scapulohumeral Rhythm and Proprioception in Patients With Rotator Cuff Tendinitis
Brief Title: Fascial Manipulation on Scapulohumeral Rhythm and Proprioception in Patients With Rotator Cuff Tendinitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/S24C08G30009 Aimen Ibrahim
Record Dates: First submitted 2025-09-25; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Rotator Cuff Tendinitis
Keywords: Fascial Manipulation; Scapulohumeral Rhythm; Proprioception; Rotator cuff tendinitis
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Fascial Manipulation technique + Conventional PT (Experimental): Fascial Manipulation in Patients with Rotator cuff tendinitis + Conventional therapy
  Interventions: Other: Fascial manipulation technique; Other: Conventional PT
- Control: Conventional PT (Active Comparator): Conventional PT including 1- hot pack (for 15 minutes)2- Periscapular exercises, a. shoulder shrug exercise (3 sets of 10 reps.) b. prone arm hangs (3 sets of 10 reps) 3- shoulder proprioception exercises a. Ball throws (30 reps) six times b. abc's on wall exercise 4- Shoulder stability exercises a. Ts Ys exercise (3 sets) b. side-lying external rotations (3 sets of 10 reps.) Total duration is 3 sessions per week for 4 consecutive weeks.
  Interventions: Other: Conventional PT

INTERVENTIONS:
Other: Fascial manipulation technique — In initially step the patient in prone position and therapist approach on the same side of the treatment limb. Use the thumb by applying the pressure on the side of the target muscle. The treatment sequence will begin with thumb gradually involve the finger. A single treatment consists of a series of specific sequences of these moves with frequent pauses 2 to 5 minutes. Treatment session duration 15-30 minutes occur 2 days per week, for 4 weeks.
  Week 1(Fascial Manipulation on the targeted muscle for 5 minutes) week 2(Fascial Manipulation on the targeted muscle for 10 minutes) week 3(Fascial Manipulation on the targeted muscle for 15 minutes) week 4 (Fascial Manipulation on the targeted muscle for 20 minutes) Conventional PT including 1- hot pack (for 15 minutes)2- Periscapular exercises, a. shoulder shrug exercise (3 sets of 10 reps.) b. prone arm hangs (3 sets of 10 reps) 3- shoulder proprioception exercises a. Ball throws (30 reps) six times
  Arms: Experimental: Fascial Manipulation technique + Conventional PT
Other: Conventional PT — Conventional PT including 1- hot pack (for 15 minutes)2- Periscapular exercises, a. shoulder shrug exercise (3 sets of 10 reps.) b. prone arm hangs (3 sets of 10 reps) 3- shoulder proprioception exercises a. Ball throws (30 reps) six times b. abc's on wall exercise 4- Shoulder stability exercises a. Ts Ys exercise (3 sets) b. side-lying external rotations (3 sets of 10 reps.) Total duration is 3 sessions per week for 4 consecutive weeks.

SUMMARY:
The aim of this randomized controlled trial is to find the effectiveness of Fascial Manipulation on Scapulohumeral Rhythm and Proprioception in Patients with Rotator cuff tendinitis

DETAILED DESCRIPTION:
Rotator cuff is a collection of four muscles (supraspinatus, infraspinatus, teres minor and subscapularis) which hold the shoulder joint and provide movement any injury to the tendon of these muscles cause rotator cuff tendinitis among all of these the supraspinatus tendon is more prone to injury because of its blood supply pattern the head of the humerus put pressure on supraspinatus tendon and hence degenerative changes started.

Rotator cuff tendinopathy typically presents with dull, aching pain around the shoulder joint, particularly over the areas of the four rotator cuff tendons. This discomfort is often aggravated by activities such as reaching overhead, reaching behind the back, lifting, or sleeping on the affected side. Pain is especially noticeable during shoulder elevation and abduction, often limiting the range of motion to less than 90° in abduction and forward flexion (anteflexion). Activities of daily living (ADLs) can become increasingly painful. The onset of pain is gradual rather than sudden and tends to persist over time The manual technique itself consists in creating localized heat by friction by using the elbow, knuckle, or fingertips on the abovementioned points. The mechanical and chemical stress effects on connective tissue are well known and a local rise in temperature could affect the ground substance of the deep fascia in these specific points. Tensional adaptation can then propagate along an entire MF sequence, diagonal, or spiral, re-establishing a physiological balance.

Fascial manipulation aims to release fascial restrictions, improve blood flow, and restore neuromuscular function. Unlike conventional treatments, FM addresses the underlying fascial adhesions that contribute to the disruption of scapulohumeral rhythm and proprioception, offering a more integrated and holistic solution to these problems. In my study, we will investigate how fascial manipulation affects proprioception and scapulohumeral rhythm in patients with rotator cuff impingement syndrome The concept that proprioception is mainly work on the mechanoreceptors which convert mechanical energy to electrical nerve impulse which give signals to central nervous system about the joint position and orientation.

* This study aims to determine if fascial manipulation can enhance the effectiveness of conventional physiotherapy by addressing myofascial restrictions that contribute to chronic tendinitis. Unlike many studies that focus on acute rotator cuff injuries, this study targets chronic cases where long-term inflammation and dysfunction persist. The research will assess long-term functional improvements rather than short-term symptom relief. While most studies focus primarily on pain reduction, this study will investigate how fascial manipulation affects scapular movement coordination and proprioceptive control, which are critical for shoulder rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Participants falling in this category would be recruited into the study.
2. Participants aged 20-45 years.
3. Gender: Male and female
4. A confirmed diagnosis of rotator cuff tendinitis based on clinical evaluation. (positive Hawkin's test, Jobe test, Empty can test, Hornblower test)
5. Persistent shoulder pain for at least 3 months.
6. Willingness to provide informed consent and adhere to the study protocol.

Exclusion Criteria:

* Participants falling in this category would be excluded from the study.

  1. History of shoulder surgery or severe structural deformities affecting the shoulder joint.
  2. Recent fracture in the upper limb.
  3. Recent dislocation in the upper limb.
  4. Uncontrolled or severe comorbidities (e.g., advanced osteoporosis, cardiovascular disease, uncontrolled diabetes).
  5. Signs or symptoms of serious underlying pathology such as infection or malignancy

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-08-30 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Lateral scapular slide test (LSST) | 4 weeks
  In the LSSTs, the distance from the inferior angle of the scapula to thoracic vertebral spinous process T8 was measured in three positions (shoulder joint 0°, 45°, and 90° abduction) using tape measures
Joint position sense test. | 4 weeks
  A laser-pointer attached to the index finger during an ART allowed measurement (mm) of JPS by measuring the distance between the target and relocated position. Participants were blindfolded and stood an arm's length (approximately 1 m) away from the wall. Whilst keeping the wrist in neutral and elbow extended, the participant actively moved to the target position (90° glenohumeral flexion), held for 5 seconds, returned their arm to their side and actively returned to the target position. A mean was calculated from three trials to provide an ART score
Goniometer | 4 weeks
  Participants will be assessed in a standardized supine position to minimize compensatory trunk or scapular movements. Bony landmarks (acromion, humeral epicondyle, mid-axillary line, olecranon process, and ulnar styloid) will be palpated for goniometer alignment. The fulcrum will be placed at the joint axis, the stationary arm aligned with the proximal reference (thorax/sternum), and the moving arm aligned with the distal segment (humerus/ulna).

CONTACTS AND LOCATIONS:
Overall Officials: Ramsha Tariq, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Life care Physiotherapy Clinic, Shahmansoor, Swabi, Swabi, Khyber Pakhunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pascoal AG, van der Helm FF, Correia PP, Carita I. Effects of different arm external loads on the scapulo-humeral rhythm. Clinical biomechanics. 2000;15:S21-S4.
- [Background] Bellotti S, Busato M, Cattaneo C, Branchini M. Effectiveness of the Fascial Manipulation Approach Associated with a Physiotherapy Program in Recurrent Shoulder Disease. Life (Basel). 2023 Jun 15;13(6):1396. doi: 10.3390/life13061396. PMID 37374178
- [Background] Day JA, Stecco C, Stecco A. Application of Fascial Manipulation technique in chronic shoulder pain--anatomical basis and clinical implications. J Bodyw Mov Ther. 2009 Apr;13(2):128-35. doi: 10.1016/j.jbmt.2008.04.044. Epub 2008 Jun 24. PMID 19329049
- [Background] Moccia D, Nackashi AA, Schilling R, Ward PJ. Fascial bundles of the infraspinatus fascia: anatomy, function, and clinical considerations. J Anat. 2016 Jan;228(1):176-83. doi: 10.1111/joa.12386. Epub 2015 Sep 25. PMID 26403802
- [Background] Szczurko O, Cooley K, Mills EJ, Zhou Q, Perri D, Seely D. Naturopathic treatment of rotator cuff tendinitis among Canadian postal workers: a randomized controlled trial. Arthritis Rheum. 2009 Aug 15;61(8):1037-45. doi: 10.1002/art.24675. PMID 19644905
- [Background] Macnab I. Rotator cuff tendinitis. Ann R Coll Surg Engl. 1973 Nov;53(5):271-87. No abstract available. PMID 4759907
- [Background] 2. Varacallo M, El Bitar Y, Mair SD. Rotator cuff tendonitis. 2018.
- [Background] 1. Rechardt M, Shiri R, Karppinen J, Jula A, Heliövaara M, Viikari-Juntura E. Lifestyle and metabolic factors in relation to shoulder pain and rotator cuff tendinitis: a population-based study. BMC musculoskeletal disorders. 2010;11:1-11.